CLINICAL TRIAL: NCT03716739
Title: Improving Quality of Life of Prostate Cancer Survivors With Androgen Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shalender Bhasin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18-733; 5R01AG060539-05 (NIH)
Record Dates: First submitted 2018-10-02; First posted 2018-10-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Active Comparator): Weekly IM administration of 100 mg testosterone cypionate for 12 weeks.
  Interventions: Drug: Testosterone Cypionate 100 MG/ML
- Control Arm (Placebo Comparator): Weekly IM administration of placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone Cypionate 100 MG/ML — 100 mg testosterone cypionate administered by intramuscular injection weekly for 12 weeks.
  Other Names: Depo-Testosterone
  Arms: Treatment Arm
Drug: Placebo — Placebo administered by intramuscular injection weekly for 12 weeks.
  Other Names: Inactive comparator
  Arms: Control Arm

SUMMARY:
The purpose of this phase II trial is to determine the efficacy and safety of testosterone replacement therapy (TRT) in improving the symptoms of androgen deficiency and health-related quality of life in men with prostate cancer who have undergone radical prostatectomy.

DETAILED DESCRIPTION:
The overall objective is to conduct a proof-of-concept double-blind, placebo-controlled, parallel group, randomized trial to determine the efficacy and safety of testosterone replacement therapy (TRT) in improving the symptoms of androgen deficiency (sexual symptoms, low energy, and physical dysfunction) and overall health-related quality of life in men with prostate cancer who have undergone radical prostatectomy for organ-localized disease (pT2,N0,M0), Gleason score < 7 (3+4), who have undetectable PSA (<0.1 ng/mL using a sensitive PSA assay) for > 2 years after radical prostatectomy, and who have androgen deficiency.

ELIGIBILITY:
Inclusion Criteria:

Men with prostate cancer, who have Stage pT2, N0, M0 lesions (confined to the gland); Combined Gleason score of 7 (3+4 elements) or less; Preoperative PSA less than 10 ng/ml; Stable and undetectable PSA level (PSA less than 0.1 ng/mL using an assay that has a functional sensitivity of 0.1 ng/mL) for at least two years after radical prostatectomy.

* Age: 40 years and older
* Presence of symptoms related to sexual dysfunction, fatigue/low vitality, or physical dysfunction.
* An average of two fasting, early morning serum testosterone levels, measured by LC-MS/MS, less than 275 mg/dL and/or free testosterone by equilibrium dialysis <60 pg/mL. middle-aged and older men with mean testosterone levels > 300 ng/dL.
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Men who have undergone radiation therapy
* Men receiving androgen deprivation therapy will be excluded.
* Hemoglobin <10 g/dL or >16.5 g/dL
* Severe untreated sleep apnea
* Allergy to sesame oil
* Uncontrolled heart failure
* Myocardial infarction, acute coronary syndrome, revascularization surgery, or stroke within 3 months
* Serum creatinine >2.5 mg/dL; ALT 3x upper limit of normal;
* Hemoglobin A1c >7.5% or diabetes requiring insulin therapy
* Body mass index (BMI) >40 kg/m2
* Untreated depression. Subjects with depression who have been on stable anti-depressant medication, or undergoing CBT for more than three months are eligible.
* Men with axis I psychiatric disorder, such as schizophrenia, will be excluded.
* Subjects who have used the following medications within the past 6 months: testosterone, DHEA, estrogens, GnRH analogs, antiandrogens, spironolactone, ketoconazole, rhGH, megestrol acetate, prednisone 20 mg daily or equivalent doses of other glucocorticoids for more than two weeks

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with a history of prostate cancer who have undergone prostatectomy.
Enrollment: 136 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
PSA Recurrence | 5-8 months
  The proportion of enrolled participations with PSA recurrence.
Change in sexual activity | 5-8 months
  Change in sexual activity is assessed by the Psychosexual Daily Questionnaire (PDQ), question 4. Subjects complete the questionnaire daily for 7 consecutive days before each visit. The PDQ covers 3 domains:1) sexual desire, enjoyment, and performance; 2) sexual activity score; and 3) mood. Sexual desire, sexual enjoyment, and mood are rated on a 7-point Likert-type scale from 0 to 7, with 0 indicating none and 7 indicating high. Activity is assessed using a checklist. Subjects record whether they had sexual daydreams; anticipation of sex; flirting; sexual interactions; and erection, masturbation, intercourse, orgasm, and ejaculation on each of the 7 days. The value is recorded as 0 (none) or 1 (any) for analysis. Weekly value is the sum of "any" responses for the week. The sexual activity score is the average of the weekly values. The score is 0 if no activity has taken place. Higher values indicate more activity and lower values indicate lower activity.

SECONDARY OUTCOMES:
Change in PSA | Baseline to 5-8 months
  Change in PSA from baseline to final assessment
Clinical Disease Recurrence | 5-8 months
  Proportion of enrolled participants with clinical disease recurrence
Change in sexual desire | 5-8 months
  Sexual desire will be assessed by DeRogatis Inventory of Sexual Function. HRQOL using the hormonal and sexual domains of the Expanded Prostate Cancer Index Composite (EPIC). Expanded Prostate Cancer Index Composite Instrument (EPIC-26) for Measuring Health-Related Quality of Life Among Prostate Cancer Survivors EPIC QOL is a 26 item questionnaire that assesses quality of life in 5 domains: urinary incontinence, urinary irritation/obstruction, bowel, sexual and vitality/hormonal domain scores.
  All domains for EPIC-26 are reported on a 0 to 100 score, with higher scores representing favorable HRQOL
Change in erectile function | 5-8 months
  Erectile function will be assessed by IIEF. The International Index of Erectile Function (IIEF) is a 15-item questionnaire that covers 4 domains of sexual function: erectile function, sexual desire, orgasmic function, and intercourse satisfaction. Each question has a potential score of 0 to 5 for a maximal score of 75 for the entire scale. Our focus in this study is on erectile function domain score, which can range from 0 to 30, lower scores indicating poor erectile function, and higher score indicating better erectile function.
Change in energy level | 5-8 months
  Energy level will be assessed using the Hypogonadism Energy Diary (HED). The total HED scale score is the sum of each of the six item weekly scores, with higher scores corresponding to greater energy level. The HED total score is linearly transformed to a scale of 0-100. Lower score indicate lower energy (or more tiredness0 and higher scores indicate more energy (less tiredness).
Change in mood | 5-8 months
  Mood and well-being will be assessed by PANAS.
Change in physical function | 5-8 months
  Physical function will be assessed by measuring stair climbing power with and without a standardized load, walking speed.
Change in self-reported physical function | 5-8 months
  Self-reported physical function will be assessed using physical function domain of MOS SF-36 (PF10)
Change in maximal voluntary strength | 5-8 months
  Maximal voluntary strength in the leg press exercise by the 1-RM method.
Change in lean body mass | 5-8 months
  Lean body mass using dual energy X-ray absorptiometry (DXA).
Change in hormone Levels | 5-8 months
  Total testosterone, DHT and estradiol will be measured using LC-MS/MS in a CDC-certified laboratory, free testosterone by equilibrium dialysis.
Change in aerobic capacity | 5-8 months
  Aerobic capacity will be assessed by measuring VO2 peak.

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts